CLINICAL TRIAL: NCT05609786
Title: Dissemination and Implementation of a Web-based Relationship Safety App, myPlanKenya, for Women at Risk for Intimate Partner Violence in Nairobi, Kenya
Acronym: myPlanKenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Ujamaa Africa (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00017456
Record Dates: First submitted 2022-11-02; First posted 2022-11-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Violence, Domestic; Violence, Sexual; Violence, Gender-Based
Keywords: Intimate Partner Violence; Relationships; Safety Planning; technology; implementation
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- myPlan Kenya (Experimental): myPlan Kenya web-based application
  Interventions: Behavioral: Personalized safety planning tool

INTERVENTIONS:
Behavioral: Personalized safety planning tool — The myPlan Kenya app is a web-based safety planning tool that is secure, private, free and personalized to the user. The app includes multiple, evidence-based modules: Strategies (safety strategies tailored to the user's needs and violence experience); Resources (referrals to local health, safety and justice resources and services); About You (questionnaires that help the user assess their relationship safety and tailor their Strategies, including My Relationship, Red Flags, My Safety, My Priorities); Understanding (knowledge sections that share information on relationships and violence, including Healthy Relationships, Harmful Beliefs About Abuse, About Violence).

SUMMARY:
This effectiveness-implementation hybrid-3 study evaluates dissemination, implementation, and effectiveness of myPlanKenya. myPlanKenya will be disseminated through formal and informal sectors. This clinical trial portion of the study enrolls women at risk for intimate partner violence (IPV) who are referred to myPlanKenya by disseminators (i.e. "end-users").

This trial aims to evaluate the effectiveness of myPlanKenya referral on resilience, health and safety among a cohort of women referred to myPlanKenya based on disclosure of IPV or assessed to have IPV related risks.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 16 or older
* Physical or sexual partner violence or relationship-based fears within the past six months; behaviorally assessed
* Living in Nairobi, Kenya with no plans to move in the next 12 months
* Access to a safe smart phone or computer (personal or shared), and comfort using it to access the myPlan Kenya app
* Literate in English or Swahili languages; confirmed by reading and completing a short passage by filling in several blanks with the appropriate words, selected from a drop-down menu.

Exclusion Criteria:

* Male
* Under age 16
* Have not experienced physical or sexual partner violence or relationship-based fears in past 6 months
* Lives outside of the study area or plans to move within the next 12 months
* Does not have access to a safe smart phone or computer, or is uncomfortable using it to access the myPlan Kenya app
* Illiterate in English or Swahili languages

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 440 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
Change in decisional conflict | Baseline, 6-month, 12-month
  12-item pre-intervention and 10-item post-intervention decisional conflict measures (specific to safety), assessed using a 5-point Likert scale (0-4). Items are scored from 0-60 pre-intervention and 0-50 post-intervention, with higher scores indicating higher lower decisional conflict and lower scores indicating higher decisional conflict.
Change in resilience as assessed by Connor-Davidson Resilience Scale | Baseline, 6-month, 12-month
  10-item Connor-Davidson Resilience Scale, which assesses resilience using a 5-point Likert scale (0-4). Items are scored from 0-40, with higher scores indicating greater resilience and lower scores indicating lower resilience.
Change in safety/IPV experience(s) as assessed by the Conflict Tactics Scale-2 | Baseline, 6-month, 12-month
  10-item adapted Conflict Tactics Scale-2 (CTS2), which assesses IPV experiences using a 3-point scale on the frequency of these experiences.
Change in help-seeking | Baseline, 6-month, 12-month
  6-item index on help-seeking, which assesses abuse disclosure and services/information received on a 2-point scale (yes/no), and the helpfulness of these disclosures and services on a 5-point Likert scale. Scale examined for fit and will be handled as individual items as needed.

SECONDARY OUTCOMES:
Change in safety strategies | Baseline, 6-month, 12-month
  5-item index on safety strategies, which assesses the use of strategies on a 2-point scale (yes/no), and the helpfulness of these strategies on a 5-point Likert scale.
Change in IPV recognition as assessed by the Abusive Behaviors Scale | Baseline, 6-month, 12-month
  7-item adapted Abusive Behaviors Scale, which assesses IPV recognition using a 5-point Likert scale (0-4). Items are scored from 0-35, with higher scores indicating greater IPV recognition and lower scores indicating lower IPV recognition.
Change in relationship intention | Baseline, 6-month, 12-month
  Single item which assesses intention for current relationship on a 4-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Decker, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Ujamaa Africa, Nairobi, Kenya